CLINICAL TRIAL: NCT03228888
Title: Effects of Ecological Rythmic-acoustic Stimulation (E-RAS) on Motor Skills in Individuals
Brief Title: Effects of Ecological Rythmic-acoustic Stimulation (E-RAS) on Motor Skills in Individuals With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Massimiliano Pau, Associate Professor, University of Cagliari
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PG/2014/17870
Record Dates: First submitted 2017-07-21; First posted 2017-07-25 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Parkinson Disease
Keywords: Rhythm; Ecological sounds; Auditory stimuli; rhythmic auditory stimulation; Parkinson's Disease; Gait; Gait analysis; Spatio-temporal parameters
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of the two groups (artificial or ecological RAS) and were evaluated in three moments: before the rehabilitative treatment (T0), at the end of the 5 week rehabilitative treatment (T5), and 3 months after the end of the treatment, namely 17 weeks after the first assessment (T17).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artificial Sounds (Experimental): Participants were provided headphones and a portable MP3 device which played a metronome tick at specified rhythm calculated as follows: a) if a patient's cadence was below the normality, the BPM of the stimulus was set at a value of 10% higher than one's own cadence; b) if a patient's cadence was below, but close to normality (less than 10% difference), the BPM of the stimulus was set at normality values; c) if a patient's cadence was above the normality, the BPM of the stimulus was set at a value equal to one's own cadence.
  Participants performed daily 30 minutes of walking assisted by the rhythmic acoustic stimuli.
  Interventions: Other: Administration of rhytmic acoustic stimuli for gait training
- Ecological Sounds (Experimental): Participants were provided headphones and a portable MP3 device which played an ecological rhythmic sound obtained by actual footsteps of human at specified rhythm calculated as follows: a) if a patient's cadence was below the normality, the BPM of the stimulus was set at a value of 10% higher than one's own cadence; b) if a patient's cadence was below, but close to normality (less than 10% difference), the BPM of the stimulus was set at normality values; c) if a patient's cadence was above the normality, the BPM of the stimulus was set at a value equal to one's own cadence.
  Participants performed daily 30 minutes of walking assisted by the rhythmic acoustic stimuli.
  Interventions: Other: Administration of rhytmic acoustic stimuli for gait training

INTERVENTIONS:
Other: Administration of rhytmic acoustic stimuli for gait training — The intervention consist in 5 weeks, 20 min/day gait training assisted by rhythmic acoustic stimuli administered using a portable MP3 player

SUMMARY:
The use of rhythmic auditory stimulation (RAS) has been proven useful in the management of gait disturbances induced by Parkinson's disease (PD). Typically, the stimuli used to provide RAS consist of metronome or music-based sounds, which are not related with the auditory experience of walking. Based on previous laboratory research, it is hypothesized that the use of ecological sounds deriving from biological motion (i.e., footstep sounds) could have a greater impact compared to artificial sounds (i.e., metronome sounds), within a rehabilitation program. In a double-blind experiment, it was investigated the effects of 5 weeks of supervised rehabilitation integrated with RAS. Thirty-two individuals affected by PD (age 68.2 ± 10.5, Hoehn and Yahr 1,5-3) were randomly assigned to one of the two conditions (artificial vs. ecological sounds). Spatio-temporal parameters of gait and clinical variables were assessed before the rehabilitation period, at its end, and after a 3-month follow-up. The results revealed that the rehabilitation program integrated with RAS had positive effects on the majority of objective and subjective measures, independently of the type of sound. However, when the two groups were examined separately, the patients assigned to the ecological RAS condition were the only who improved both in terms of cadence and gait speed. Overall, the hypothesized greater effect of the ecological sounds compared to artificial sounds was only partially supported by data.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of PD according to the UK Brain Bank criteria;
* ability to walk independently;
* absence of relevant hearing impairments which could prevent the correct perception of the auditory cues;
* absence of significant cognitive impairment (i.e., Mini-Mental Status Examination (MMSE) > 24; Frontal Assessment Battery (FAB) > 13);
* absence of psychiatric or severe systemic illnesses;
* mild-to-moderate disability assessed by means of the modified Hoehn and Yahr (H&Y) staging scale (1,5 ≤ H&Y ≤ 3);
* no engagement in any rehabilitative program in the 3 months before the beginning of the study

Exclusion Criteria:

-

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Walking speed | 5 weeks
  Walking speed calculated on a 10 m path using motion-capture system

SECONDARY OUTCOMES:
Hip Flexion-extension | 5 weeks
  Angle of flexion-extension of hip joint during a gait cycle
Knee Flexion-extension | 5 weeks
  Angle of flexion-extension of knee joint during a gait cycle
Ankle Dorsi- Plantar-flexion | 5 weeks
  Angle of dorsi- plantar-flexion of ankle joint during a gait cycle
GPS | 5 weeks
  Gait Profile Score (synthetic index of deviation from a physiologic gait pattern)

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital "G. Brotzu", Cagliari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Murgia M, Pili R, Corona F, Sors F, Agostini TA, Bernardis P, Casula C, Cossu G, Guicciardi M, Pau M. The Use of Footstep Sounds as Rhythmic Auditory Stimulation for Gait Rehabilitation in Parkinson's Disease: A Randomized Controlled Trial. Front Neurol. 2018 May 24;9:348. doi: 10.3389/fneur.2018.00348. eCollection 2018. PMID 29910764